CLINICAL TRIAL: NCT04442477
Title: Neurodevelopment at 5.5 Years of Age in Children Who Received Infant Formula With Enriched Protein Fractions
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: 6027-2
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Cognitive Ability, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Enriched Protein Fractions: This group was given Infant formula with enriched protein fractions
  Interventions: Dietary Supplement: Enriched Protein Fractions
- Active Comparator: Protein Fractions: This group was given Infant formula with protein fractions
  Interventions: Dietary Supplement: Protein Fraction

INTERVENTIONS:
Dietary Supplement: Enriched Protein Fractions — Enriched protein fractions
  Groups: Experimental: Enriched Protein Fractions
Dietary Supplement: Protein Fraction — Protein fractions
  Groups: Active Comparator: Protein Fractions

SUMMARY:
This is a follow-up study of a multi-center, double-blind, randomized, controlled, parallel-designed, prospective trial and is intended to evaluate neurodevelopment at 5.5 years of age and health outcomes through 5.5 years of age in participants who received one of two staged study formulas through one year of age.

ELIGIBILITY:
Inclusion Criteria:

* Participant who previously consumed study formula through one year of age in MJN Project 6027
* 5.5 years of age (i.e. when child turns 5 years and 6 months old ± 2 months) at Visit 1
* Signed informed consent obtained for child's participation in the study

Exclusion Criteria:

* No exclusion criteria

Ages: 64 Months to 68 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants who previously consumed study formula through one year of age in MJN Project 6027.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Wechsler Preschool & Primary Scale of Intelligence™ (Fourth Edition; WPPSI™-IV) | At 5.5 years of age

SECONDARY OUTCOMES:
Dimensional Change Card Sort (DCCS) | At 5.5 years of age
Stroop Task | At 5.5 years of age
Functional Near Infrared Spectroscopy (fNIRS) | At 5.5 years of age
Child Behavior Checklist (CBCL) | At 5.5 years of age
Body weight | At 5.5 years of age
Body height | At 5.5 year of age
Health history outcomes | At 5.5 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, Principal Investigator — Shanghai Children's Medical Center; Steven Wu, M.D., Study Director — Mead Johnson/RB
Locations (1):
- Fuyang Fifth People's Hospital, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colombo J, Harris CL, Wampler JL, Zhuang W, Shaddy DJ, Liu BY, Wu SS. Improved Neurodevelopmental Outcomes at 5.5 Years of Age in Children Who Received Bovine Milk Fat Globule Membrane and Lactoferrin in Infant Formula Through 12 Months: A Randomized Controlled Trial. J Pediatr. 2023 Oct;261:113483. doi: 10.1016/j.jpeds.2023.113483. Epub 2023 May 14. PMID 37192722